CLINICAL TRIAL: NCT06312306
Title: Effect of Transcranial Direct Current Stimulation Versus Pilates Based Core Stability Training on Balance and Gait in Stroke Patients
Brief Title: Transcranial Direct Current Stimulation vs Pilates Core Training in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aisha Mohamed Khaled Ahmed Saleh, M.Sc. in Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDCS vs pilates in stroke
Record Dates: First submitted 2024-02-24; First posted 2024-03-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: stroke; tDCS; core training; pilates; gait; balance
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial direct current stimulation (tDCS) group (Experimental): Anodal tDCS applied using a DC stimulator
  Interventions: Device: transcranial direct current stimulation; Other: conventional physiotherapy program
- pilates based core training group (Experimental): The Pilates training program will last 30 min per session. The selected exercises will be given to all patients and progressed week-wise
  Interventions: Other: Pilates based core training; Other: conventional physiotherapy program
- control group (Active Comparator): Will receive conventional physiotherapy program
  Interventions: Other: conventional physiotherapy program

INTERVENTIONS:
Device: transcranial direct current stimulation — Anodal tDCS applied using a direct current stimulator and two saline-soaked electrodes. The anode electrodes will be positioned approximately 2 cm anterior to Cz according to the International 10/20 EEG System. The cathode will be positioned over the inion. Stimulation intensity will be at 2.0 milliampere (as suggested to achieve excitation in the lower limb motor cortex areas)
  Arms: Transcranial direct current stimulation (tDCS) group
Other: Pilates based core training — The Pilates training program will last 30 min per session, Each action in the training will be repeated eight times these actions are at beginner level, considering the characteristics of stroke patients. The selected exercises will be given to all patients and progressed week-wise.
  Arms: pilates based core training group
Other: conventional physiotherapy program — Conventional physiotherapy program:
  * Stretching Slow sustained stretching of spastic muscles (generally hip flexors and adductors, knee extensors or flexors and ankle plantar flexors)
  * Strengthening Abdominals, lumbar spine extensors, hip flexors, extensors and abductors, knee extensors and flexors and ankle dorsi flexors
  * Gait training In level surface and in stairs

SUMMARY:
The goal of this clinical trial is to compare the effects of transcranial direct current stimulation and pilates based core stability training on gait and balance in stroke patients. The main question[s] it aims to answer are:

* is there an effect of transcranial direct current stimulation and pilates based core training on gait and balance
* Is there a significant effect of tDCS over Pilates-based core training

Participants will be assigned to three groups:

* Group 1: will receive 18 sessions(3 sessions/week 20 minutes each) of anodal tDCS in addition to conventional physical therapy exercises
* Group 2: Will receive 18 Pilates exercise sessions over a period of 6 weeks (3 sessions / week) in addition to conventional physical therapy exercises.
* Group 3: Will receive conventional physiotherapy program

Researchers will compare the transcranial direct current stimulation group with the pilates exercise group to see if one of them is superior to the other on balance and gait.

DETAILED DESCRIPTION:
The ultimate goal for rehabilitation is to enhance functional performance in various essential real life activities. There is a need for a more effective, cost-efficient treatments for balance and gait in stroke patients. Many studies have reported that Pilates exercise has positive effects in development of muscular strength, endurance, flexibility, and in prevention of falls in elderly population and in orthopedic rehabilitation. However, there are only a few studies available with Pilates as intervention in neurological conditions such as multiple sclerosis, Parkinson's disease and stroke. This study aims to evaluate the efficacy of Pilates exercise on balance, in post stroke survivors and thereby provide an evidence for further studies in neurological conditions. Transcranial direct current stimulation(tDCS) is a promising noninvasive neuromodulatory intervention that aims to maximize recovery of function after stroke. There are numerous arguments to suggest that tDCS may become interesting tools to promote gait and balance improvement in stroke patients. The ability of these techniques to modulate cortical excitability was demonstrated. However, very few study has examined the effect of stimulating the SMA with tDCS on balance and gait performance. Motor learning is crucial in human daily life, both throughout the lifespan as well as for the recovery from a variety of neurological diseases. The ability of both exercise such as pilates and non invasive neuromodulation such as tDCS to modulate cortical excitability and therefore enhance motor learning has been demonstrated. Therefore, the aim of this study is to compare the effect of a Pilates-based core training program and tDCS over the supplementary motor area on balance and gait in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with either hemorrhagic or ischemic stroke for the first time, with an onset of more than eight weeks
* Their age should be 50-60 years old.
* Patients of a minor (1-4) to moderate (5-15) national institutes of health stroke scale (NIHSS) score.
* Sufficient cognitive ability to participate, as indicated by Mini-mental state examination score of 21 or higher.
* ambulatory before stroke
* ability to stand or walk with or without assistance
* mild to moderate spasticity (MAS scale less than grade 3)
* hemodynamically stable

Exclusion Criteria:

* History of seizures.
* Patients with Any medical metal devices incompatible with transcranial direct current stimulation (e.g. pacemaker).
* Bi-hemispheric or multifocal stroke.
* any other neurological pathology affecting balance (cerebellar or brain stem lesions, impaired vision, visual field defect or hemineglect)
* Premorbid neurological impairment prior to onset of stroke.
* Co-morbidities impairing the motor function such as fracture or deformity.
* Medically unstable.
* Mental and cognitive impairment.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Gait kinematics | 6 weeks
  Gait video will be recorded by a high-definition digital camera, and analysis will be done by Kinovea 2D motion analysis software
The Biodex Balance System | 6 weeks
  The Biodex Balance System (BBS; Biodex Inc.) will be used to assess postural stability.
  The BBS measures, in degrees, the tilt about each axis during dynamic conditions and calculates a medial-lateral stability index, anterior-posterior stability index, and an overall stability index.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | 6 weeks
  Quality of life was measured using the SIS Version 3.0 which is a 59 item self report scale designed to measure a person's perspective of the effect of stroke on quality of life. The SIS assesses eight domains: strength, hand function, activity of daily living, mobility, communication, emotion, memory and thinking, and participation. Each item was rated on a five point ordinal scale where five was "not difficult at all" to one which was "extremely difficult". Summative scores are generated for each domain and can range from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Saleh, Principal Investigator — Cairo University; Hussein Shaker, Professor, Study Director — cairo univeristy; Ebtesam Fahmy, Professor, Study Director — Cairo University; Mohamed Helayel, lecturer, Study Chair — cairo univeristy
Locations (1):
- Faculty of physical therpay cairo university, Dokki, Giza Governorate, Egypt